CLINICAL TRIAL: NCT00793299
Title: Burden of Cancer in Children: A Pilot Study to Investigate the Impact and Content of Video Illness Narratives
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Barbara Asselin, Pediatrics, Hematology Oncology, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RSRB00025699
Record Dates: First submitted 2008-11-18; First posted 2008-11-19 (Estimated); Last update posted 2015-04-27 (Estimated); Status verified 2015-04

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Video Illness Narrative (Experimental): single arm pilot study
  Interventions: Behavioral: Video Illness Narrative

INTERVENTIONS:
Behavioral: Video Illness Narrative — video

SUMMARY:
In order to gain a greater understanding of the full experience of children with life-threatening illness, this study will provide video cameras to ten to fifteen 10-18 years olds in active treatment for cancer, and instruct them to make video illness narratives over the course of 1-3 months. The narratives will be studied as an intervention; each of the participants will be administered a measure of physical symptoms (the Memorial Symptom Assessment scale 10-18) and a measure of self-esteem (the Rosenberg Self-Esteem Scale). The video narratives will also be analyzed for content by theme in order to understand the participants' experiences in their own words. Our hypothesis is that these narratives will provide insight into the lives of children with cancer, increase their self-esteem, and decrease symptom distress, and improve communication between patients and their doctors.

DETAILED DESCRIPTION:
In addition to the above outcome measures:

The video narratives will also be analyzed for content by theme in order to understand the participants' experiences in their own words.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with cancer
* Age 10-18
* In active treatment for cancer
* Followed at the Strong Memorial Hospital/Golisano Children's Hospital

Exclusion Criteria:

* Non-English Speaker
* Cognitively impaired so as to make data collection difficult

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 11 (Actual)
Dates: Start 2008-11; Primary Completion 2009-06 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Memorial Symptom Assessment Scale | 3 months

SECONDARY OUTCOMES:
Rosenberg Self Esteem Scale | 3 mopnths

CONTACTS AND LOCATIONS:
Overall Officials: Emily Hahn, BA, Principal Investigator — Medical Student; Barbara Asselin, MD, Principal Investigator — Associate Professor
Locations (1):
- University of Rochester School of Medicine and Dentistry, Golisano Children's Hospital at Strong, Rochester, New York, United States